CLINICAL TRIAL: NCT04162080
Title: Observational Study in Kayak Polo Athletes.
Brief Title: Kayak Polo Athletes
Acronym: KYAth
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, Principal Investigator, University of Valencia
Other Study IDs: ID0028
Record Dates: First submitted 2019-11-10; First posted 2019-11-14 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Athletes
Keywords: kayak polo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kayak polo (KP) is a sport that, as a breviary, can be defined as the union between water polo and canoeing. The objective of this study is to compare anthropometric parameters, joint assessment, strength and functional capacity between two groups of KP players from the Valencian Community. The sample will be divided into a Sub21 group and a Senior group. Anthropometric variables (body mass index [BMI], percentage of fat mass, waist - hip index [CHF], body perimeters ...), shoulder assessment (Range of movement in rotations, Scapular Dyskinesis Test [SDT]) will be assessed. glenohumeral instability ...), hip assessment (modified Thomas test), strength (Hand Grip Strength test and upper limb thrust), lower limb power (Counter Movement Jump [CMJ]) and functional capacity (1 'push-ups for limbs upper and 1 'Sit-to-Stand test for lower limbs).

ELIGIBILITY:
Inclusion Criteria:

* kayak polo athletes

Exclusion Criteria:

* other sports
* current injuries the previous 6 months

Ages: 16 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: Observational cross-sectional study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Weight and percentage of fat mass | 1 day
  A scale - bioimpedaniometer model Tanita BF350 Anazyliser body composition will be used. Through acoustic bioimpedance, the four sensors of this scale that come into contact with the soles of the feet serve to assess the body composition of the individual, once the data on: size, age and sex have been entered.
Skin fold | 1 day
  An 842-SK-001 polymer pyrometer of the Quirumed brand will be used. This one has an accuracy of 2mm and will be used for the measurement of skin folds of adipose tissue. Specifically, the tricipital fatty fold (PGT) will be measured
Shoulder ROM | 1 day
  To obtain the ROM in shoulder rotations, a conventional analog polymer goniometer of the Saehan brand Grip model will be used, with an accuracy of 2 degrees. External rotation (RE) and internal rotation (RI) of the dominant upper limb will be assessed.

SECONDARY OUTCOMES:
Scapular dyskinesia | 1 day
  To assess the scapular dyskinesia, one of the most expanded tests in terms of the evaluation of the scapular kinematics will be used: the SDT. It consists of an observational assessment: the subject to study will be placed in standing position with his back to the examiner and performed between 5-10 shoulder abductions and the same number of shoulder flexions bilaterally (Figure 2-1) with a light load on each hand; The examiner is positioned so that he can observe the scapular kinematics without interference. Once done, it is classified as: absence of scapular dyskinesia or presence of scapular dyskinesia (subtle or obvious). It is a test with moderate inter-examiner reliability and high intra-examiner reliability.
Glenohumeral apprehension test | 1 day
  The glenohumeral apprehension test (IGH) is used to evaluate IGH. This test consisted of placing the subject in standing position with 90º shoulder abduction and 90º elbow flexion passively. From this position, the examiner performs a posteroanterior displacement of the head of the humerus. The test is positive if the examinee shows signs of apprehension (running away from the posture, rotating to avoid displacement of the humeral head, ...) or indicating subjective sensation of instability
Impingement subacromial (SAPS) | 1 day
  Based on the work of Diercks R et al and concluding that a single test is not sufficient to identify the presence of shoulder pathology, the combination of different tests is chosen to make a more reliable diagnosis for SAPS.
Shortening in hip flexion | 1 day
  To assess the possible shortening of the hip flexor muscles, the modified Thomas test with pelvic stabilization will be used, since without external stabilization authors have determined that it is easy to obtain false positives.
  The subject under examination is placed supine on the stretcher with approximately 3/4 of the lower limbs outside the stretcher. From that position a cinch is placed that stabilizes at the level of the anterior superior iliac spines, it is instructed to bring the knees to the chest and hold one of them with the hands. The leg to be evaluated is the one that is extended and the presence of passive hip flexion or not is assessed.
  Two measurements are made per lower limb, the test was positive if the subject unintentionally is unable to keep the thigh of the leg to be tested in contact with the stretcher.
Clamping force in upper limbs | 1 day
  It is used for the test of maximum grip strength in upper limb (HGS). With the subject in sitting position, with elbow flexion of 90, he is instructed to perform the maximum clamping force on the hydraulic hand dynamometer, so as to alter as little as possible the initial posture.
  The dynamometer is of the analog hydraulic type of the Jamar model SP-5030J1, adjusting the grip according to the size of the subject's hand. This gives us a value that ranged from 0 to 90kg.
Thrust force in upper limbs | 1 day
  To assess the thrust force of the upper limbs, an estimate of the maximum load (in kilograms) capable of moving a single vertical position in a flat bench press is performed, that is, the 1RM assessment is performed during the press exercise. hde banking. 1RM, Refers to the maximum load (in kg) that is able to move a subject in a given movement, which defines the maximum force of a subject for a particular exercise.
Movement Jump (CMJ) or Countermovement Jump | 1 day
  It is done by starting with the subject from an upright position with the hands on the iliac crests. From this position the subject performs a flexion quickly followed by an extension of lower limbs which triggers the jump. At no time does the subject help himself with the upper limbs to apply inertia. This assessment is done by using the iPhone application "My Jump 2". First, a profile is created in the application for each subject where it is introduced: body weight, lower limb length measured with tape measure from the trochanter to fingertips with maximum plantar flexion and height from the ground to the trochanter with lower limbs in half-squat with both knees at 90 degrees of flexion. The smartphone and the subject are placed following the scheme shown in Figure 2-3. The subject performs the CMJ and the smartphone by using the slow motion the exact height (in centimeters) of the jump made in a valid way is calculated
Functional capacity in lower limbs | 1 day
  The functional capacity of lower limbs is established by the 1 minute Sit-to-stand test. This assessment consists of getting up and sitting from a chair (45 cm high) as many times as possible for a minute. Two series are performed and the average of both measurements is obtained.
  This objectification, validated by several authors, offers us a value that is directly proportional to the functional capacity. That is, greater number of repetitions means greater functional capacity of lower limbs.
Functional ability in upper limbs | 1 day
  The functional capacity of upper limbs is established by the 1 minute Push-up test. Push-ups are performed with 4 supports on the floor: both feet and both hands. From this plate position flexion - extension of upper limbs is performed as many times as possible for one minute.
  This objectification, validated by several authors, offers us a value that is directly proportional to the functional capacity. That is, greater number of repetitions means greater functional capacity of lower limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, Dr, Principal Investigator — Faculty of Physiotherapy. University of Valencia
Locations (2):
- Spain (2):
  - Gemma Espí, Valencia
  - Gemma v. Espí López, Valencia

IPD SHARING:
Plan to Share IPD: No